CLINICAL TRIAL: NCT01197586
Title: Evaluation of Surfactant Protein B in the Differential Diagnostics of Dyspnea
Status: Completed | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Principal Investigator, Joachim Saur, Principal Investigator, Universitätsmedizin Mannheim
Other Study IDs: 2010_spb_ma
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Dyspnea; Cardiac Disease; Pulmonary Disease
Keywords: surfactant protein B; differential diagnostics
MeSH Terms: conditions — Dyspnea; Heart Diseases; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Establishing new biochemical markers in the differential diagnostics and risk stratification in heterogeneous patient collectives is becoming more and more important. The markers should be objective, reliable, reproducible, quick and cost effective as well as specific and sensitive. Concerning the differential diagnostics of "dyspnea", NT-pro-BNP plays the most important role for the evaluation of a cardiac origin. However, a corresponding biochemical marker for pulmonary stress is lacking. The aim of the study at hand therefore was the evaluation of surfactant protein B in the differential diagnostics of pulmonary and cardiac diseases.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting with dyspnea and giving informed consent

Exclusion Criteria:

* outpatients
* lack or doubt of legal competence
* indication for mechanical ventilation
* pregnancy
* palliative patients
* CPAP/LTOT
* BMI > 30 kg/m2
* sepsis
* anemia
* dialysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients presenting with the symptom "dyspnea" in a university hospital emergency room
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Surfactant protein B serum levels | Days 1, 3 and 7

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Saur, MD, Principal Investigator — Universitätsmedizin Mannheim
Locations (1):
- Universitaetsmedizin Mannheim, Mannheim, Germany